CLINICAL TRIAL: NCT04365907
Title: Enhanced Extraction Technique of Omarigliptin From Human Plasma: Applied to Biological Samples From Healthy Human Volunteers
Brief Title: Omarigliptin in Four Healthy Egyptian Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Bassam Mahfouz Ayoub, Associate Professor in Analytical Chemistry Department,, British University In Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CDRD-3
Record Dates: First submitted 2020-04-17; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omarigliptin 12.5 mg (Experimental): Drug: Omarigliptin 12.5 mg Once weekly new anti-diabetic drug approved only in Japan Other Name: Zafatek tablets
  Interventions: Drug: Zafatek tablets

INTERVENTIONS:
Drug: Zafatek tablets — Once weekly new anti-diabetic drug approved only in Japan

SUMMARY:
The proposed study will consider the LC-MS/MS quantitative determination of Omarigliptin after administration to four Egyptian volunteers. The main aim of the study is to confirm that the developed LC-MS/MS method is applicable for the bio-assay of the drug in the actual biological samples at the time of Cmax (nearly about 1.5 hours). The design of the study is open labeled, one treatment, one period, single dose study. The concentration of the drugs after 1.5 h will be determined in healthy human subjects according to the ethical regulations of World Medical Association Declaration of Helsinki (October 1996) and the International Conference of Harmonisation Tripartite Guideline for Good Clinical Practice. Written informed consent was provided (attached and signed by the four volunteers) in order to be approved by the ethics committee of the Faculty of Pharmacy, The British University in Egypt. The good health of the human subjects was confirmed by a complete medical history and physical examination. Samples from four, healthy, adult, male, smoking, Egyptian volunteers (age: 23-37 years, Average weight: 81.6 kg, Average BMI: 30.4) will be collected at 1.5 h, to be transferred to heparinized centrifuge tubes in order to be analyzed by LC-MS/MS study (developed & validated) after single oral dose administration of one Marizev® tablet nominally containing 12.5 mg of Omarigliptin (first arm as 4 volunteers). The blood samples (1 mL of each sample) will be centrifuged at 3000 rpm for 5 minutes, 100 µL of the plasma will be separated and spiked with the internal standard working solution and then the sample preparation and LC-MS/MS determination will be applied. Blood glucose level will be determined for all volunteers at different time intervals to monitor any hypoglycemic effect to ensure their safety all over the study. The study will be conducted as per FDA guidelines & the evaluation of safety of the study will be based on monitoring of blood glucose level, vital signs, pulse rate, monitoring of adverse events, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Must be able to swallow tablets

Exclusion Criteria:

* Insulin dependent diabetes
* Type-2 diabetes
* Hospitalized within 1 week

Ages: 23 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-28 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration (nMol/L) after 1.5 hours | 1.5 hours
  Only one determination of human plasma concentration (nM/L) of omarigliptin will be determined after 1.5 hours for the current investigation.

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, El-Sherouk, Egypt

IPD SHARING:
Plan to Share IPD: Undecided